CLINICAL TRIAL: NCT05794594
Title: 3D Printed Personalized Extendable Prosthesis Replacement for Limb Preservation in Children With Osteosarcoma: a Preliminary Study
Brief Title: 3D Printed Personalized Extendable Prosthesis
Status: Completed | Type: Observational
Sponsor: Yuxi Su (Other)
Responsible Party: Sponsor-Investigator, Yuxi Su, Children's Hospital of Chongqing Medical University, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: CHChongqingMU-2
Record Dates: First submitted 2023-03-18; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Osteosarcoma in Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3D printed: 3D printed personalized extendable prosthesis replacement for limb preservation in children with osteosarcoma
  Interventions: Device: 3D printed personalized extendable prosthesis
- amputation: patients had undergone amputation of the limbs

INTERVENTIONS:
Device: 3D printed personalized extendable prosthesis — 3D printed personalized extendable prosthesis replacement for limb preservation in children
  Groups: 3D printed

SUMMARY:
The goal of this type of observational study is to investigate the preliminary effect of 3D printed personalized extendable prosthesis replacement on limb salvage in children with osteosarcoma. The main question it aims to answer is:

Is 3D printed personalized extendable prosthesis replacement has a good outcome in limb salvage pediatric osteosarcoma？

DETAILED DESCRIPTION:
Osteosarcoma is one of the most common primary malignant bone tumors in children and adolescents. In this study, the investigators try to investigate the preliminary effect of 3D printed personalized extendable prosthesis replacement on limb salvage in children with osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* tumors of the extremities, with moderate soft-tissue invasion
* the neurovascular bundle is not invaded, and the tumor can be excised totally
* no metastatic lesions or metastases can be cured

Exclusion Criteria:

* recurrent tumors
* poorly differentiated tumors
* poor soft-tissue conditions
* neurovascular invasion around tumors
* ineffective chemotherapy with metastasis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children with osteosarcoma undergoing prosthesis replacement or limb amputation were admitted to our hospital
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Recurrence | 7years
  Osteosarcoma recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Yuxi Su, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided